CLINICAL TRIAL: NCT07324122
Title: EVALUATION OF THE EFFECT OF RECRUITMENT MANEUVER ON POSTOPERATIVE ATELECTASIS IN LAPAROSCOPIC CHOLECYSTECTOMY SURGERY USING LUS (LUG ULTRASOUND SCALE)
Brief Title: Effect of Recruitment Maneuver on Postoperative Atelectasis Assessed by Lung Ultrasound in Laparoscopic Cholecystectomy
Acronym: LUNG USG SCORE
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FSMTRHLUS; 2025-KAEK-43 (Other: ISTANBUL PROVINCIAL DIRECTORATE OF HEALTH KOŞUYOLU HIGH SPECIALIZATION EDUCATION AND CLINICAL RESEARCH ETHICS COMMITTEE)
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Perioperative Atelectasis During Laparoscopic Cholecystectomy
Keywords: recruitment, lung ultrasound score, laparoscopic cholecystectomy, atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No biological samples will be taken from the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Extubation Recruitment Group: Patients undergoing laparoscopic cholecystectomy in whom a standardized alveolar recruitment maneuver is applied prior to extubation, with perioperative lung aeration evaluated using lung ultrasound score.
- Standard Ventilation Group: Patients undergoing laparoscopic cholecystectomy managed with standard mechanical ventilation without application of a recruitment maneuver. Lung aeration is evaluated perioperatively using lung ultrasound scoring.

SUMMARY:
This study is an observational clinical investigation designed to evaluate perioperative lung aeration in adult patients undergoing elective laparoscopic cholecystectomy under general anesthesia. The primary objective is to assess lung status using lung ultrasound in patients aged 18 to 65 years.

A total of 80 volunteer participants will be enrolled. Lung aeration will be evaluated using lung ultrasound scoring before and after surgery. Patient demographic characteristics, medical history, intraoperative airway pressure values, and perioperative lung ultrasound scores will be recorded for analysis.

This study is conducted solely for research purposes and does not involve any drug intervention. All patients will receive standard perioperative care as determined by their attending anesthesiologist and surgical team, with no deviation from routine clinical practice. Participation is voluntary, and patients may withdraw from the study at any time without affecting their medical care.

DETAILED DESCRIPTION:
Perioperative atelectasis is a frequent consequence of general anesthesia and represents a major contributor to postoperative pulmonary complications. Anesthesia-induced loss of functional residual capacity, impaired diaphragmatic movement, and altered ventilation-perfusion matching predispose dependent lung regions to alveolar collapse. These effects are further amplified during laparoscopic surgery due to pneumoperitoneum-induced increases in intra-abdominal pressure, patient positioning, and the routine use of high fractions of inspired oxygen. Even in patients without preexisting pulmonary disease, these factors may result in clinically significant atelectasis during and after surgery.

Laparoscopic cholecystectomy is one of the most commonly performed minimally invasive surgical procedures and serves as a standardized clinical model to investigate perioperative respiratory strategies. Pneumoperitoneum and reverse Trendelenburg positioning during this procedure lead to cephalad displacement of the diaphragm, reduced lung compliance, and regional ventilation heterogeneity, thereby increasing the risk of perioperative atelectasis.

Alveolar recruitment maneuvers are ventilation strategies aimed at reopening collapsed alveoli by temporarily increasing transpulmonary pressure. When applied appropriately, recruitment maneuvers may improve lung aeration, enhance oxygenation, and increase respiratory system compliance. Several studies have demonstrated the beneficial effects of recruitment maneuvers during laparoscopic surgery; however, the optimal timing of these maneuvers remains controversial. The period immediately before extubation is particularly vulnerable to lung derecruitment, and applying a recruitment maneuver at this time may help restore lung aeration and reduce early postoperative atelectasis.

Lung ultrasound has emerged as a reliable, noninvasive, and bedside imaging modality for the assessment of lung aeration. The Lung Ultrasound Score (LUS) allows semi-quantitative evaluation of aeration loss by systematically examining predefined thoracic regions. LUS has been validated against computed tomography and has demonstrated high sensitivity in detecting perioperative atelectasis, making it well suited for use in the intraoperative and immediate postoperative period.

In this prospective clinical study, adult patients scheduled for elective laparoscopic cholecystectomy under general anesthesia will be evaluated to determine the effect of an alveolar recruitment maneuver applied immediately before extubation on perioperative atelectasis. Lung aeration will be assessed using lung ultrasound at predefined time points, and changes in the Lung Ultrasound Score will be used as the primary indicator of atelectasis. Secondary outcomes will include oxygenation parameters and basic respiratory variables.

This study aims to provide objective ultrasound-based evidence regarding the effectiveness of pre-extubation recruitment maneuvers in reducing perioperative atelectasis. The findings may contribute to the optimization of lung-protective ventilation strategies in routine anesthetic practice and support the integration of lung ultrasound into perioperative respiratory monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective laparoscopic cholecystectomy under general anesthesia
* Age between 18 and 65 years
* Body mass index (BMI) < 30 kg/m²
* American Society of Anesthesiologists (ASA) physical status classification I-III
* Provision of written informed consent

Exclusion Criteria:

* Refusal to participate in the study
* Emergency surgical procedures
* Body mass index (BMI) ≥ 30 kg/m²
* American Society of Anesthesiologists (ASA) physical status classification IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 65 years who are scheduled to undergo elective laparoscopic cholecystectomy under general anesthesia. Eligible participants have a body mass index below 30 kg/m² and are classified as American Society of Anesthesiologists (ASA) physical status I-III. All participants provide written informed consent prior to enrollment. Patients undergoing emergency surgery or with significant comorbidities requiring ASA physical status IV are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
change in lung ultrasound score (LUS) | From preoperative baseline to 30 minutes postoperatively
  Perioperative change in lung aeration assessed by lung ultrasound score using a standardized 12-quadrant examination. LUS values obtained preoperatively and at 30 minutes postoperatively will be compared between the recruitment maneuver group and the standard ventilation group.

CONTACTS AND LOCATIONS:
Overall Officials: doga meric yukselen, MD, Study Director — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL; elif acar deger, MD, Study Chair — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL; oznur demiroluk, MD, Study Chair — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL; arzu yildirim ar, MD, Study Chair — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL; arsen gungor ay, MD, Study Director — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL; cansu ofluoglu, MD, Principal Investigator — ISTANBUL PROVINCIAL HEALTH DIRECTORATE FATIH SULTAN MEHMET TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Istanbul Provincial Health Directorate Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Result] Liu Y, Wang J, Geng Y, Zhang Y, Su H, Yang Y. The effect of ultrasound-guided lung recruitment maneuvers on atelectasis in lung-healthy patients undergoing laparoscopic gynecologic surgery: a randomized controlled trial. BMC Anesthesiol. 2022 Jul 1;22(1):200. doi: 10.1186/s12871-022-01742-1. PMID 35778701
- [Result] Kim BR, Lee S, Bae H, Lee M, Bahk JH, Yoon S. Lung ultrasound score to determine the effect of fraction inspired oxygen during alveolar recruitment on absorption atelectasis in laparoscopic surgery: a randomized controlled trial. BMC Anesthesiol. 2020 Jul 18;20(1):173. doi: 10.1186/s12871-020-01090-y. PMID 32682397